CLINICAL TRIAL: NCT05715775
Title: Enlightenment of Robotic Gastrectomy From 527 Patients With Gastric Cancer in the Minimally Invasive Era: 5 Years of Optimizing Surgical Performance in a High-volume Center
Brief Title: Learning Curve and Optimization of Robotic Gastrectomy
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director of gastric surgery, Fujian Medical University
Other Study IDs: RGLC-01
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
we explore the learning curve and the impact of technique optimization on surgical outcomes and the first to construct a referenceable learning phase for performing robotic gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Case inclusion criteria: (1) patients with pathologically confirmed gastric adenocarcinoma; (2) no distant metastases; and (3) R0 resection was performed.

Exclusion Criteria:

* Case exclusion criteria: (1) the presence of distant metastases was found ; (2) preoperative neoadjuvant chemotherapy was administered; and (3) clinical information was incomplete.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 527 patients who underwent RG between August 2016 and June 2021.
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The LN dissection rate | 36 months
  The LN dissection rate was defined as the number of the LN station was examined divided by the total number of retrieval LN station.

SECONDARY OUTCOMES:
LN noncompliance | 30 days
  LN noncompliance was defined as the absence of LNs from more than 1 LN station.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xue Z, Lu J, Lin J, Xu KX, Xu BB, Wu D, Zheng HL, Xie JW, Wang JB, Lin JX, Chen QY, Li P, Huang CM, Zheng CH. Enlightenment of robotic gastrectomy from 527 patients with gastric cancer in the minimally invasive era: 5 years of optimizing surgical performance in a high-volume center - a retrospective cohort study. Int J Surg. 2024 Sep 1;110(9):5605-5614. doi: 10.1097/JS9.0000000000001652. PMID 38775618